CLINICAL TRIAL: NCT00117208
Title: A Cross-Over Comparative Study of Inhaled Mannitol, Alone and in Combination With Daily rhDNase, in Children With Cystic Fibrosis
Brief Title: Comparison of Inhaled Mannitol and rhDNase in Children With Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Syntara (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DPM-CF-203
Record Dates: First submitted 2005-06-30; First posted 2005-07-04 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-01

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Mannitol; dornase alfa

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: mannitol
- 2 (Active Comparator): DNase daily for 12 weeks
  Interventions: Drug: Dornase alpha
- 3 (Other): combination
  Interventions: Drug: mannitol + pulmozyme

INTERVENTIONS:
Drug: mannitol — 400mg BD for 12 weeks
  Arms: 1
Drug: mannitol + pulmozyme — combination
  Arms: 3
Drug: Dornase alpha — 2.5mg daily for 2 weeks
  Other Names: rhDNase, pulmozyme
  Arms: 2

SUMMARY:
The purpose of this study is to determine the medium term efficacy and safety profile of inhaled mannitol, on its own and also as an additional therapy to rhDNase (pulmozyme). In particular, we will assess the impact on: lung function; airway inflammation; sputum microbiology; exacerbations; quality of life; adverse events; exercise tolerance; total costs of hospital and community care; and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Known diagnosis of cystic fibrosis (sweat test or genotype)
* Of either gender
* Aged between 8 and 18 years
* Have a baseline FEV1 of <70% of the predicted normal value
* Currently taking rhDNase for at least 4 weeks

Exclusion Criteria:

* Currently active asthma, uncontrolled hypertension, colonised with Burkholderia cepacia or MRSA
* Listed for transplantation
* Known intolerance to mannitol, rhDNase or bronchodilators

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2005-11; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
FEV1 after 12 weeks of each of the following treatment regimens: *mannitol only *rhDNase only *mannitol + rhDNase | 12 weeks

SECONDARY OUTCOMES:
to compare mannitol to rhDNase on FVC | 12 weeks
to assess whether the effects of mannitol are additive to rhDNase | 12 weeks
to demonstrate that mannitol does not cause deterioration in airway inflammation | 12 weeks
to assess whether mannitol reduces the bacterial load in the lung | 12 weeks
to assess whether the effects of mannitol are beneficial to quality of life | 12 weeks
to assess whether mannitol, or mannitol + rhDNase are cost-effective compared to rhDNase alone | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Bush, FRCPCH, Principal Investigator — Royal Brompton and Harefiled NHS Trust; Colin Wallis, FRCPCH, Principal Investigator — Great Ormond Street Hospital for Children NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Great Ormond Hospital for Children, London
  - Royal Brompton Hospital, London

REFERENCES:
- [Background] Suri R, Metcalfe C, Lees B, Grieve R, Flather M, Normand C, Thompson S, Bush A, Wallis C. Comparison of hypertonic saline and alternate-day or daily recombinant human deoxyribonuclease in children with cystic fibrosis: a randomised trial. Lancet. 2001 Oct 20;358(9290):1316-21. doi: 10.1016/S0140-6736(01)06412-1. PMID 11684212
- [Background] Robinson M, Daviskas E, Eberl S, Baker J, Chan HK, Anderson SD, Bye PT. The effect of inhaled mannitol on bronchial mucus clearance in cystic fibrosis patients: a pilot study. Eur Respir J. 1999 Sep;14(3):678-85. doi: 10.1034/j.1399-3003.1999.14c30.x. PMID 10543292
- [Background] Daviskas E, Anderson SD, Brannan JD, Chan HK, Eberl S, Bautovich G. Inhalation of dry-powder mannitol increases mucociliary clearance. Eur Respir J. 1997 Nov;10(11):2449-54. doi: 10.1183/09031936.97.10112449. PMID 9426077
- [Background] Daviskas E, Anderson SD, Eberl S, Chan HK, Bautovich G. Inhalation of dry powder mannitol improves clearance of mucus in patients with bronchiectasis. Am J Respir Crit Care Med. 1999 Jun;159(6):1843-8. doi: 10.1164/ajrccm.159.6.9809074. PMID 10351929
- [Background] Daviskas E, Anderson SD, Eberl S, Chan HK, Young IH. The 24-h effect of mannitol on the clearance of mucus in patients with bronchiectasis. Chest. 2001 Feb;119(2):414-21. doi: 10.1378/chest.119.2.414. PMID 11171717
- [Background] Daviskas E, Anderson SD, Gomes K, Briffa P, Cochrane B, Chan HK, Young IH, Rubin BK. Inhaled mannitol for the treatment of mucociliary dysfunction in patients with bronchiectasis: effect on lung function, health status and sputum. Respirology. 2005 Jan;10(1):46-56. doi: 10.1111/j.1440-1843.2005.00659.x. PMID 15691238
- [Result] Minasian C, Wallis C, Metcalfe C, Bush A. Comparison of inhaled mannitol, daily rhDNase and a combination of both in children with cystic fibrosis: a randomised trial. Thorax. 2010 Jan;65(1):51-6. doi: 10.1136/thx.2009.116970. Epub 2009 Dec 8. PMID 19996349
- [Result] Minasian C, Wallis C, Metcalfe C, Bush A. Bronchial provocation testing with dry powder mannitol in children with cystic fibrosis. Pediatr Pulmonol. 2008 Nov;43(11):1078-1084. doi: 10.1002/ppul.20903. PMID 18972410
- [Derived] Yang C, Montgomery M. Dornase alfa for cystic fibrosis. Cochrane Database Syst Rev. 2021 Mar 18;3(3):CD001127. doi: 10.1002/14651858.CD001127.pub5. PMID 33735508
- [Derived] Enderby B, Doull I. Hypertonic saline inhalation in cystic fibrosis--salt in the wound, or sweet success? Arch Dis Child. 2007 Mar;92(3):195-6. doi: 10.1136/adc.2006.094979. PMID 17337677